CLINICAL TRIAL: NCT06920563
Title: Remote Postpartum Blood Pressure Monitoring and Cardiovascular Education to Reduce Emergency Department Visits, Re-admissions and Adverse Cardiovascular Outcomes in Hypertensive Disorder of Pregnancy
Brief Title: Remote Postpartum Blood Pressure Monitoring and Cardiovascular Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.192
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Pre-Eclampsia; Complicating Pregnancy; Gestational Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Hypertension, Pregnancy-Induced | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This group will watch an education video, receive text message updates, and have their blood pressure medications titrated to a lower BP goal.
  Interventions: Other: Video; Other: Text Reminder; Other: Blood pressure threshold
- Control (No Intervention): This group will receive usual post partum care from their obstetrician

INTERVENTIONS:
Other: Video — Those in the intervention arm will watch a short educational video.
  Arms: Intervention
Other: Text Reminder — Those in the intervention group will receive regular text message reminders to check their blood pressures
  Arms: Intervention
Other: Blood pressure threshold — Those in the intervention group will have a lower blood pressure threshold to titrate their BP medications towards
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if patient education and regular text reminders are a feasible intervention to engage patients and reduce post partum hypertension. The main questions it aims to answer are:

Is a structured postpartum remote blood pressure monitoring intervention with education and individualized medication initiation/adjustment follow-up by televisit feasible? Does a structured program reduce the occurrence of postpartum hypertension, ED visits, hospital readmissions, and adverse outcomes?

Participants will:

View an educational video on HDP post-delivery Receive 1-2 times daily text messages for 6 weeks postpartum Have their blood pressure medications adjusted to lower targets post partum

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Postpartum status.
3. Experience new-onset hypertension during pregnancy.
4. Enrollment in Connected MOM.
5. Ability to provide informed consent.
6. Establish medical care within the Ochsner System to facilitate data collection.

Exclusion Criteria:

1. History of preeclampsia or gestational hypertension during previous pregnancy
2. History of chronic hypertension
3. History of coronary artery disease (myocardial infarction, coronary stent placement, coronary artery bypass grafting, spontaneous coronary artery dissection)
4. History of ischemic CVA
5. History of Congestive heart failure
6. Renal dysfunction
7. Liver dysfunction
8. Left ventricular dysfunction
9. Congenital heart disease
10. Still birth at delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Engagement | 6 weeks
  Engagement will be defined by frequency of use: number of remote BP measurements ascertained during the 6 week postpartum period.
Acceptability | 6 weeks
  Post program survey questions using 5-item Likert response scale at 6 weeks postpartum
Duration of Participation | 6 weeks
  Duration of participation is defined by the last day of recorded remote BP measurement

SECONDARY OUTCOMES:
Post partum Blood pressure | 1 year
  Proportion of patients with BP <130/80 at 6 weeks Mean SBP, DBP at 6 weeks, 6 months, 1 year postpartum
Number of ED visits | 1 year
  Number of ED visits recorded after discharge from her delivery encounter over the following year.
Severe Maternal Morbidity | 1 year
  Incidence of death, postpartum stroke, congestive heart failure, myocardial infarction, eclampsia
Number of Inpatient re-admissions | 1 year
  Number of inpatient re-admissions over the following year after discharge from delivery encounter
Post partum visit follow up | 6 weeks
  Proportion of 4-6 week postpartum follow up visit attendance with OB provider

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Baptist, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mitro SD, Hedderson M, Xu F, Forquer H, Baker JM, Kuzniewicz MW, Greenberg M. Risk of postpartum readmission after hypertensive disorder of pregnancy and variation by discharge antihypertensive medication prescription. Am J Obstet Gynecol. 2024 Oct;231(4):456.e1-456.e13. doi: 10.1016/j.ajog.2024.01.015. Epub 2024 Jan 25. PMID 38280432
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Cairns AE, Tucker KL, Leeson P, Mackillop LH, Santos M, Velardo C, Salvi D, Mort S, Mollison J, Tarassenko L, McManus RJ; SNAP-HT Investigators. Self-Management of Postnatal Hypertension: The SNAP-HT Trial. Hypertension. 2018 Aug;72(2):425-432. doi: 10.1161/HYPERTENSIONAHA.118.10911. Epub 2018 Jul 2. PMID 29967037
- [Background] Kitt JA, Fox RL, Cairns AE, Mollison J, Burchert HH, Kenworthy Y, McCourt A, Suriano K, Lewandowski AJ, Mackillop L, Tucker KL, McManus RJ, Leeson P. Short-Term Postpartum Blood Pressure Self-Management and Long-Term Blood Pressure Control: A Randomized Controlled Trial. Hypertension. 2021 Aug;78(2):469-479. doi: 10.1161/HYPERTENSIONAHA.120.17101. Epub 2021 Jun 28. PMID 34176288
- [Background] Hauspurg A, Lemon LS, Quinn BA, Binstock A, Larkin J, Beigi RH, Watson AR, Simhan HN. A Postpartum Remote Hypertension Monitoring Protocol Implemented at the Hospital Level. Obstet Gynecol. 2019 Oct;134(4):685-691. doi: 10.1097/AOG.0000000000003479. PMID 31503166
- [Background] Mujic E, Parker SE, Nelson KP, O'Brien M, Chestnut IA, Abrams J, Yarrington CD. Implementation of a Cell-Enabled Remote Blood Pressure Monitoring Program During the Postpartum Period at a Safety-Net Hospital. J Am Heart Assoc. 2024 Jul 2;13(13):e034031. doi: 10.1161/JAHA.123.034031. Epub 2024 Jun 27. PMID 38934890
- [Background] Bateman BT, Schumacher HC, Bushnell CD, Pile-Spellman J, Simpson LL, Sacco RL, Berman MF. Intracerebral hemorrhage in pregnancy: frequency, risk factors, and outcome. Neurology. 2006 Aug 8;67(3):424-9. doi: 10.1212/01.wnl.0000228277.84760.a2. PMID 16894102
- [Background] Jeng JS, Tang SC, Yip PK. Stroke in women of reproductive age: comparison between stroke related and unrelated to pregnancy. J Neurol Sci. 2004 Jun 15;221(1-2):25-9. doi: 10.1016/j.jns.2004.03.006. PMID 15178209
- [Background] Bushnell C, Chireau M. Preeclampsia and Stroke: Risks during and after Pregnancy. Stroke Res Treat. 2011 Jan 20;2011:858134. doi: 10.4061/2011/858134. PMID 21331165
- [Background] Benschop L, Duvekot JJ, Versmissen J, van Broekhoven V, Steegers EAP, Roeters van Lennep JE. Blood Pressure Profile 1 Year After Severe Preeclampsia. Hypertension. 2018 Mar;71(3):491-498. doi: 10.1161/HYPERTENSIONAHA.117.10338. PMID 29437895
- [Background] Honigberg MC, Zekavat SM, Aragam K, Klarin D, Bhatt DL, Scott NS, Peloso GM, Natarajan P. Long-Term Cardiovascular Risk in Women With Hypertension During Pregnancy. J Am Coll Cardiol. 2019 Dec 3;74(22):2743-2754. doi: 10.1016/j.jacc.2019.09.052. Epub 2019 Nov 11. PMID 31727424
- [Background] Haug EB, Horn J, Markovitz AR, Fraser A, Klykken B, Dalen H, Vatten LJ, Romundstad PR, Rich-Edwards JW, Asvold BO. Association of Conventional Cardiovascular Risk Factors With Cardiovascular Disease After Hypertensive Disorders of Pregnancy: Analysis of the Nord-Trondelag Health Study. JAMA Cardiol. 2019 Jul 1;4(7):628-635. doi: 10.1001/jamacardio.2019.1746. PMID 31188397
- [Background] Wu P, Haththotuwa R, Kwok CS, Babu A, Kotronias RA, Rushton C, Zaman A, Fryer AA, Kadam U, Chew-Graham CA, Mamas MA. Preeclampsia and Future Cardiovascular Health: A Systematic Review and Meta-Analysis. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003497. doi: 10.1161/CIRCOUTCOMES.116.003497. Epub 2017 Feb 22. PMID 28228456
- [Background] Fasanya HO, Hsiao CJ, Armstrong-Sylvester KR, Beal SG. A Critical Review on the Use of Race in Understanding Racial Disparities in Preeclampsia. J Appl Lab Med. 2021 Jan 12;6(1):247-256. doi: 10.1093/jalm/jfaa149. PMID 33227139
- [Background] Ouyang P, Sharma G. The Potential for Pregnancy Heart Teams to Reduce Maternal Mortality in Women With Cardiovascular Disease. J Am Coll Cardiol. 2020 Nov 3;76(18):2114-2116. doi: 10.1016/j.jacc.2020.09.007. No abstract available. PMID 33121719
- [Background] Gad MM, Elgendy IY, Mahmoud AN, Saad AM, Isogai T, Sande Mathias I, Misbah Rameez R, Chahine J, Jneid H, Kapadia SR. Disparities in Cardiovascular Disease Outcomes Among Pregnant and Post-Partum Women. J Am Heart Assoc. 2021 Jan 5;10(1):e017832. doi: 10.1161/JAHA.120.017832. Epub 2020 Dec 16. PMID 33322915
- [Background] Rana S, Lemoine E, Granger JP, Karumanchi SA. Preeclampsia: Pathophysiology, Challenges, and Perspectives. Circ Res. 2019 Mar 29;124(7):1094-1112. doi: 10.1161/CIRCRESAHA.118.313276. PMID 30920918
- [Background] Croke L. Gestational Hypertension and Preeclampsia: A Practice Bulletin from ACOG. Am Fam Physician. 2019 Nov 15;100(10):649-650. No abstract available. PMID 31730305